CLINICAL TRIAL: NCT04960163
Title: Incidence and Predictors of Bleeding Diathesis Development Due to DIC in Cirrhosis and ACLF Patients Undergoing CRRT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-ACLF-08
Record Dates: First submitted 2021-06-17; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention
  Other Names: This is an observational Study

SUMMARY:
ACLF and cirrhotic patient have deranged coagulation parameters and this coagulation parameters altered when this group of patients undergoing dialysis because of renal failure. this group of patients is also high risk of sepsis. Most common organ involved during sepsis leading to organ failure is renal. So, all this cascade increases the risk of bleeding as well as coagulation failure. Currently there are no studies evaluation the coagulation status in patients with cirrhosis undergoing dialysis. Further there are no studies evaluating the utility of these global tests of coagulation as a guide to judicious blood transfusion in these patients to prevent bleeding. Further there are no studies comparing the two different modalities of assessment.

DETAILED DESCRIPTION:
METHODOLOGY Aim: The incidence and predictors of bleeding diathesis development due to DIC in cirrhosis and ACLF patients undergoing CRRT

Primary Objective:

Primary: Development of bleeding diathesis within 3 days [ e.g-bleeding/ooze from access sites, GI bleeding (blood in ryles tube, hematemesis's, melena, bleeding PR), bleed form ET tube site, bleed form nose/mouth or any other site]

Secondary Objective:

1. Assess the following factors as predictors of bleeding diathesis within 3 days:

   * Severity of liver disease: CTP, MELD, MELD-Na, APACHE, SOFA, AARC, lactate, ammonia, [baseline and degree of change ,12 hrly,24 ,48 and 72 Hrly]
   * Presence and severity of AKI, HE [baseline and degree of change 12 hrly,24,48,72 or at the detection of bleeding]
   * Presence and severity of infections/sepsis [baseline and degree of change 12 hrly or at the detection of bleeding]
   * Complement levels (C3/C4) [baseline and degree of change at day 3 or at the detection of bleeding]
   * Following test of coagulation system [baseline and degree of change 12 hrly,24,48,72 hrly and at the detection of bleeding [ Platelets counts (manual), PT(INR), Prothrombin index, aPTT, Factor VIII/vWF , Fibrinogen, d-Dimer, FDP, DIC score)
   * ROTEM (EXTEM,FIBTEM,APTEM,INTEM)
   * Type and dose vasopressors (NA, vaso, Terlipressin, somat, phenylep)
   * Hemodynamic parameters [pulse, BP, Lung water, SVV, SVR, CO/CI] optional
   * CRRT parameters [type of dialysate, membrane, flow,]
2. Survival by day 7

Study Population: Patients with cirrhosis or ACLF undergoing CRRT.

Study Design: A prospective study.

Study Period

* The study will be conducted on patients admitted to Department of Hepatology from May 2021 to Aug 2021 at ILBS, New Delhi
* Study group will comprise of patients with cirrhosis undergoing dialysis.

Sample size with Justification: There are no previous study to determine the bleeding risk in ACLF or cirrhotic patient undergoing CRRT therapy so this is the pilot study so taking first 40 patients.

Intervention: There are no intervention arm. its prospective trial.

Monitoring and assessment: Investigator will be monitoring any bleeding epiosdes during the CRRT and in case there are any bleeding risk the coagulation factors based upon ROTEM and correct the coagulation abnormalties will be done.

Statistical Analysis:

* All variables shall be expressed in median (range)
* Variables will be compared by Mann- Whitney U test
* For Categorical variables we will use Chi-Square or Fisher's test
* Survival analysis will be done using cox-proportional regression analysis

Actuarial probability of survival shall be calculated by Kaplan- Meier graph and compared by log- rank test.

Adverse Effects: increase risk of bleeding during CRRT

Stopping rule of Study: in case of bleeding not controlled with coagulation correction or patient become hemodynamically unstable , negative consent for the further course of treatment then study will be stopped .

Expected outcome of the project-.

Primary end points:

Incidence of dialysis related bleeding in first 24 hours

Secondary end points:

1. To assess correlation of ROTEM abnormalities with risk of clinically significant bleeding
2. To assess the need and volume of FFP, Cryoprecipitate, platelet and packed red blood cell transfusion based on ROTEM pre- and post-procedure
3. Incidence of transfusion associated lung injury and circulatory overload in both groups at 24 hours
4. Incidence of infections (Time frame first 24 hours)
5. Incidence of infections and bleeding in first 7 days
6. Duration of hospital or ICU stay in both groups
7. 7 day mortality.

ROTEM would be done pre-procedure to assess the coagulation status for all patients enrolled and subsequently post procedure and in case of bleeding, after transfusion at 12 hours and 24 hours, 48 and 72 hours respectively. Other standard blood tests would be done including record of mean arterial pressures, CBC, KFT, LFT, PT/INR, arterial ammonia, lactate, serum procalcitonin as required. In case of presence or absence of active bleed FFPs, Cryoprecipitate, platelets will be transfused depending upon the coagulation parameters as assessed by ROTEM .

ELIGIBILITY:
Inclusion Criteria:

- Consecutive patients with cirrhosis or ACLF undergoing their first session of dialysis

Exclusion Criteria:

1. Age <12 or > 75 years
2. Hepatocellular Carcinoma
3. Recent history of blood product transfusion in the last 7 days
4. History of antiplatelets, antifibrinolytics or antithrombotics
5. Active untreated Sepsis/DIC
6. Any evidence of active bleed secondary to coagulopathy
7. Pregnancy
8. Comorbidities associated with poor outcome (Extrahepatic neoplasia, severe cardiopulmonary disease defined by a New York Heart Association score >3, or oxygen/steroid-dependent chronic obstructive pulmonary disease )
9. Refusal to participate in the study.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cirrhosis or ACLF undergoing CRRT.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dialysis related bleeding in first 24 hours | 24 hours

SECONDARY OUTCOMES:
To assess correlation of ROTEM abnormalities with risk of clinically significant bleeding | 24 hours
To assess the volume of FFP pre- and post-procedure | 24 hours
To assess the volume of Cryoprecipitate pre- and post-procedure | 24 hours
To assess the volume of platelet pre- and post-procedure | 24 hours
To assess the volume of packed red blood cell transfusion based on ROTEM pre- and post-procedure | 24 hours
Incidence of transfusion associated lung injury and circulatory overload in both groups at 24 hours | 24 hours
Incidence of infections | 24 hours
Incidence of infections | 7 days
Incidence of bleeding | 7 days
Duration of Intensive Care Unit or hospital | 7 days
Mortality | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No